CLINICAL TRIAL: NCT06926608
Title: Actívatexto: Advancing Smoking Cessation and Physical Activity Among Latinos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, Francisco Cartujano, MD, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009837; R01MD019748 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Smoking; Smoking Cessation; Physical Inactivity
MeSH Terms: conditions — Smoking; Smoking Cessation; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Actívatexto (Experimental): Actívatexto is a mobile intervention that promotes both smoking cessation and physical activity. Actívatexto integrates four components: 1) a text messaging program that promotes both smoking cessation and physical activity, 2) wearable devices to monitor physical activity, 3) smoking cessation pharmacotherapy (i.e., nicotine replacement therapies), and 4) an online dashboard where the research team manages participants' incoming and outgoing data from both the text messaging program and wearable devices.
  Interventions: Behavioral: Actívatexto
- Decídetexto (Active Comparator): Decídetexto is a mobile intervention that solely promotes smoking cessation. Decídetexto integrates three components: 1) a text messaging program that solely promotes smoking cessation, 2) smoking cessation pharmacotherapy (i.e., nicotine replacement therapies), and 3) an online dashboard where the research team manages participants' incoming and outgoing data from the text messaging program.
  Interventions: Behavioral: Decídetexto

INTERVENTIONS:
Behavioral: Actívatexto — Actívatexto is a mobile intervention that promotes both smoking cessation and physical activity. Actívatexto integrates four components: 1) a text messaging program that promotes both smoking cessation and physical activity, 2) wearable devices to monitor physical activity, 3) smoking cessation pharmacotherapy (i.e., nicotine replacement therapies), and 4) an online dashboard where the research team manages participants' incoming and outgoing data from both the text messaging program and wearable devices.
  Arms: Actívatexto
Behavioral: Decídetexto — Decídetexto is a mobile intervention that solely promotes smoking cessation. Decídetexto integrates three components: 1) a text messaging program that solely promotes smoking cessation, 2) smoking cessation pharmacotherapy (i.e., nicotine replacement therapies), and 3) an online dashboard where the research team manages participants' incoming and outgoing data from the text messaging program.
  Arms: Decídetexto

SUMMARY:
The purpose of this randomized controlled trial is to assess the efficacy of Actívatexto (Aim 1) and the mediators of the presumed treatment effect (Aim 2) among Latino adults who smoke. Actívatexto is a mobile intervention that integrates four components: 1) a text messaging program that promotes both smoking cessation and physical activity, 2) wearable devices to monitor physical activity, 3) smoking cessation pharmacotherapy [i.e., nicotine replacement therapies (NRT)], and 4) an online dashboard where the research team manages participants' incoming and outgoing data from both the text messaging program and wearable devices.

DETAILED DESCRIPTION:
We will conduct a two-arm randomized controlled trial among Latinos who smoke and do not meet the recommended levels of physical activity (N=408). Participants will be recruited via community-based efforts and randomly assigned in a 1:1 ratio to Actívatexto (a mobile intervention that promotes both smoking cessation and physical activity) or Decídetexto (a mobile intervention that solely promotes smoking cessation). All participants will be provided with nicotine replacement therapies and a Fitbit Versa 4 device. Participants in both groups will complete a baseline assessment at enrollment and follow-up assessments at Months 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic and/or Latino
* Know how to read and speak English and/or Spanish
* Be ≥ 18 years of age
* Not meet the recommended levels of physical activity (150 minutes of moderate to vigorous physical activity)
* Smoke cigarettes at least 3 days per week
* Be interested in quitting smoking in the next 30 days
* Have a cellphone with text messaging capability
* Know how to utilize text messages
* Be willing to wear a wearable device daily to monitor physical activity
* Be willing to complete all study visits

Exclusion Criteria:

* Use of tobacco products other than cigarettes in the past 30 days (including e-cigarettes)
* Being pregnant or breastfeeding
* Plan to move from their current residence in the next six months
* Another household member enrolled in the study
* Unable to become more physically active or engage in a fitness appraisal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with cotinine verified 7-day point prevalence abstinence | Month 6
  Cotinine levels ≤15 ng/mL in saliva

SECONDARY OUTCOMES:
Percent of participants with self-reported 7-day point prevalence abstinence | Month 6
  No cigarettes, "not even a puff", in the past 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No